CLINICAL TRIAL: NCT00938899
Title: Phase I, Double Blind, Randomized, Placebo-controlled Trial in Healthy Subjects to Examine the Safety, Tolerability and Pharmacokinetics of Increasing Oral Doses of TMC435350 After Single and Repeated Dosing, Followed by an Open Label Repeated Dosing Session in 6 HCV genotype1 Infected Patients.
Brief Title: TMC435350-TiDP16-C101 - A Study to Examine the Safety, Tolerability and Pharmacokinetics of Increasing Oral Doses of TMC435350 After Single and Repeated Dosing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Compound Development Team Leader, Tibotec Pharmaceuticals Limited, Ireland
Other Study IDs: CR012610
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Hepatitis C
Keywords: TMC435350-TiDP16-C101; TMC435350-C101; TMC435350; HCV
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir

INTERVENTIONS:
Drug: TMC435350; Placebo

SUMMARY:
The purpose of this study is to examine the safety, tolerability and pharmacokinetics of increasing oral doses of TMC435350 after single and repeated dosing, followed by an open label repeated dosing session in 6 HCV genotype1 infected patients.

DETAILED DESCRIPTION:
This trial is a randomized, double blind, placebo-controlled trial to determine the safety, tolerability and pharmacokinetics of TMC435350 after single and multiple oral doses taken by healthy non-Hepatitis C Virus infected (non-HCV) participants, followed by an open label repeated doses taken by 6 HCV-genotype 1 infected participants (non-placebo controlled). The single dose escalation part of the trial will consist of 6 sessions (Sessions Ia to VIa) and will include 2 panels of 9 healthy non-HCV infected participants each (Panels 1 and 2). The dose of the test drug will be consecutively escalated. Doses of 50 mg, 100 mg, 200 mg, 400 mg, 800 mg and 1200 mg of TMC435350 or placebo will be administered as a single oral administration alternating over the 2 panels. In each session, 6 participants will receive active treatment and 3 participants will receive placebo after a breakfast. The treatment schedule will ensure that over 3 sessions each particpant will receive active treatment twice and placebo once. There is a washout period of at least 10 days between consecutive TMC435350 or placebo dosings within each panel. Participants of Panel 1 will have an additional session to investigate food effect: a single dose of TMC435350 will be tested in fasted conditions (Session VIIa). Food effect will be investigated for the 200 mg dose in Panel 1, unless the the available concentration of the drug in the blood and safety data from previous sessions prove unnecessary. Multiple dosing will be started when Sessions Ia (single dose of 50 mg), IIa (single dose of 100 mg) and IIIa (single dose of 200 mg) are found to be safe and tolerable. The multiple dose escalation part of the trial will consist of 4 consecutive sessions (Sessions Ib to IVb) in 4 panels of 9 healthy non-HCV infected participants each (Panels 3, 4, 5 and 6). In each session, 6 participants will receive active treatment and 3 participants will receive placebo. TMC435350 or placebo will be administered during 5 consecutive days. As a potential food effect is not yet known, administration will be after a meal. Treatment is anticipated to be twice daily with doses of 50 mg, 100 mg, 200 mg and 400 mg. The available concentration of the drug in the blood will be determined up to 72 hours after the first dose, in case a single dose of TMC435350 is given (in Sessions Ia to VIIa and, if performed, Session VIIIa). In case of multiple dosing (in Sessions Ib to IVb), full pharmacokinetic profiles of TMC435350 will be determined for the first dosage interval (e.g. up to 24 hours after the first dose for a b.i.d. regimen) and up to 72 hours after the last dose. Safety and tolerability will be evaluated continuously and documented (safety report), with 24-hours interim PK data after the last dose, before stepping up to the next dose and between each session. After completion of the healthy participant sessions, an open label session (Ic) in HCV genotype 1 infected participant will be added. The trial population (Panel 7) will include 6 male or female, non-responder HCV-genotype 1 infected participants with an HCV viral load of at least 50000 IU/mL. These participants will be treated as Panel 7 with follow-up visits, after the 5 day dosing period. One dose regimen will be selected which was shown to be safe in healthy participants and as close as possible to a maximum tolerated dose, which will be administered for 5 days. In addition to drug safety and PK parameters, viral loads will be determined in plasma.

ELIGIBILITY:
Inclusion Criteria:

- Healthy participants must be non-smokers, normal weight, normal ECG, healthy on the basis of a medical evaluation, physical examination, medical history, ECG, vital signs, and laboratory results

* HCV patients must be of normal weight, normal ECG, chronic genotype 1 HCV infection, non-responders or relapsers to previous treatment regimens and have a HCV viral load at least 50000 IU/mL plasma at screening.

Exclusion Criteria:

* Patients with history of cardiac disease, HIV-1 or HIV-2 test
* Women of childbearing potential
* History or evidence of abuse of alcohol, barbiturate, amphetamine, recreational or narcotic drug use, hepatitis A, B or C infection
* Positive urine drug test
* Any active or underlying disease
* History of drug allergy or hypersensitivity
* Participation in an investigational trial within 30 days prior to the first intake of study medication
* Recent donation of blood
* Abnormal laboratory values
* HCV patients with cardiac disease, co-infections with HIV-1, HIV-2 or liver infection other than HCV
* Women of childbearing potential
* Participants not agreeing to use a reliable birth control method until last trial visit
* Drug abuse
* Cardiovascular, hepatic or renal disease, diabetes, epilepsy, skin or psychiatric disease
* Enrolled in another clinical trial for 90 days prior to screening
* Evidence of Child Pugh B or C liver disease
* Having received a polymerase or protease inhibitor treatment during the last 6 months
* Abnormal laboratory values

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2007-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Determine the safety, tolerability and pharmacokinetics of TMC435350 after single oral doses from 50 mg up to 1200 mg and after 5 days of dosing from 50 mg up to 400 mg or up to Multiple dosing. | Pharmacokinetics and safety at time of drug intake until 72hour after the drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Limited Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- [Derived] Reesink HW, Fanning GC, Farha KA, Weegink C, Van Vliet A, Van 't Klooster G, Lenz O, Aharchi F, Marien K, Van Remoortere P, de Kock H, Broeckaert F, Meyvisch P, Van Beirendonck E, Simmen K, Verloes R. Rapid HCV-RNA decline with once daily TMC435: a phase I study in healthy volunteers and hepatitis C patients. Gastroenterology. 2010 Mar;138(3):913-21. doi: 10.1053/j.gastro.2009.10.033. Epub 2009 Oct 21. PMID 19852962
- See also: Phase I, double blind, randomized, placebo-controlled trial in healthy subjects to examine safety, tolerability, PK of increasing single and repeating oral doses of TMC435, followed by an open label repeated dosing session in 6 HCV G1 infected patients. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=1008&filename=CR012610_CSR.pdf